CLINICAL TRIAL: NCT01269736
Title: Implementation of Practice Standards for ECG Monitoring
Acronym: PULSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 0711003292; R01HL081642 (NIH)
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-06

CONDITIONS: Cardiovascular Disease
Keywords: electrocardiographic monitoring; arrhythmia; myocardial ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac; Myocardial Ischemia | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Online ECG monitoring education program and strategies to implement and sustain change for nurses
  Interventions: Behavioral: Education
- Control (No Intervention): Usual in-service education for nurses

INTERVENTIONS:
Behavioral: Education — Online ECG monitoring education program and strategies to implement and sustain change for nurses
  Arms: Education

SUMMARY:
The purpose of this study is to test the effect of implementing new practice standards for electrocardiographic (ECG) monitoring on nurses' knowledge and skills, quality of care, and patient outcomes. The investigators hypothesize that increased knowledge and skills of nurses will lead to enhanced quality of care, which will result in improved outcomes for patients.

DETAILED DESCRIPTION:
Despite advances in hospital electrocardiographic (ECG) monitoring technology, monitoring practices are inconsistent and often inadequate. The investigators recently published practice standards for ECG monitoring. The primary purpose of this 5-year multisite randomized clinical trial is to test the effect of implementing these standards on nurses' knowledge and skills, quality of care, and patient outcomes. The investigators expect that increased knowledge and skills of nurses will lead to enhanced quality of care, which will result in improved outcomes for patients. Units serving cardiac patients in 17 hospitals will participate. Hospitals will be randomized to the experimental or control group after baseline measures of knowledge and skills, quality of care, and patient outcomes are obtained. The intervention will include ECG monitoring education and strategies to implement and sustain change. The online education will include 4 modules: essentials of ECG monitoring, arrhythmia monitoring, ischemia monitoring, and QT interval monitoring. The strategies to implement and sustain change in the clinical area include reinforcement of education, incentives, and the designation of "champions" on each unit who will actively promote the implementation of the practice standards.

ELIGIBILITY:
Inclusion Criteria:

* Nurses (and monitor technicians): All nurses (and monitor technicians) working on participating units serving patients with cardiac disease
* Patients: All patients cared for on participating units

Exclusion Criteria:

* Nurses (and monitor technicians): No nurses (or monitor technicians) will be excluded
* Patients: No patients on the participating units will be excluded, even if their primary diagnosis is not cardiac

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92057 (Actual)
Dates: Start 2008-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Funk, PhD, RN, Principal Investigator — Yale University School of Nursing
Locations (16):
- United States (14):
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Maine Medical Center, Portland, Maine
  - Baystate Medical Center, Springfield, Massachusetts
  - United Hospital, Saint Paul, Minnesota
  - Erie County Medical Center, Buffalo, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Seton Medical Center, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Meriter Heart Hospital, Madison, Wisconsin
- University of Ottawa Heart Institute, Ottawa, Canada, Ottawa, Ontario, Canada
- Hong Kong Sanatorium & Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Funk M, Rose L, Fennie K. Challenges of an Internet-based education intervention in a randomized clinical trial in critical care. AACN Adv Crit Care. 2010 Oct-Dec;21(4):376-9. doi: 10.1097/NCI.0b013e3181e6765d. PMID 21045576
- [Result] Funk M, Winkler CG, May JL, Stephens K, Fennie KP, Rose LL, Turkman YE, Drew BJ. Unnecessary arrhythmia monitoring and underutilization of ischemia and QT interval monitoring in current clinical practice: baseline results of the Practical Use of the Latest Standards for Electrocardiography trial. J Electrocardiol. 2010 Nov-Dec;43(6):542-7. doi: 10.1016/j.jelectrocard.2010.07.018. Epub 2010 Sep 15. PMID 20832819
- [Result] Funk M, Fennie KP, Stephens KE, May JL, Winkler CG, Drew BJ; PULSE Site Investigators. Association of Implementation of Practice Standards for Electrocardiographic Monitoring With Nurses' Knowledge, Quality of Care, and Patient Outcomes: Findings From the Practical Use of the Latest Standards of Electrocardiography (PULSE) Trial. Circ Cardiovasc Qual Outcomes. 2017 Feb;10(2):e003132. doi: 10.1161/CIRCOUTCOMES.116.003132. PMID 28174175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In addition to the nurses and patients consented in each hospital, 95,884 hospital admission records were reviewed for patient outcomes, representing 84,392 unique patients from 13 hospitals.
Pre-assignment Details: Hospitals were the unit of randomization, nurses received ECG education in each hospital. Outcomes were assessed in nurses and the patients cared for on the participating units.
Units Other Than Participants: Hospitals
Groups:
- Online ECG Education: The intervention consisted of an online ECG monitoring education program (9 mo) and strategies to implement and sustain change in practice (6 mo). Data were collected from both groups at time 2 after group 1 received the intervention. Final data collection occurred at time 3 after group 2 received the intervention. Data collection time points were 15 mo apart.
- Standard Care Then Online ECG Monitoring: Hospitals were randomized to administer usual in-service education for nurses for 15 months, then received an online ECG monitoring education program (9 mo) and strategies to implement and sustain change in practice (6 mo). Data were collected from both groups at time 2 after group 1 received the intervention. Final data collection occurred at time 3 after group 2 received the intervention. Data collection time points were 15 mo apart.
Period: Nurses' Knowledge Assessments
Arm/Group | Online ECG Education | Standard Care Then Online ECG Monitoring
Started | 1585; 9 Hospitals (873 unique nurses were assessed at 9 hospitals at the initiation of the study.) | 1428; 8 Hospitals (866 unique nurses were assessed at 8 hospitals at the initiation of the study.)
Baseline Assessment | 873; 9 Hospitals (873 unique nurses, assessed at 9 hospitals.) | 866; 8 Hospitals (866 unique nurses, assessed at 8 hospitals.)
15 Months Assessment | 1108; 9 Hospitals (1108 unique nurses, assessed at 9 hospitals.) | 782; 8 Hospitals (866 unique nurses, assessed at 8 hospitals.)
30 Months Assessment | 741; 8 Hospitals (741 unique nurses, assessed at 8 hospitals.) | 926; 8 Hospitals (926 unique nurses, assessed at 8 hospitals.)
Completed | 1585; 8 Hospitals (1585 unique nurses assessed overall (at any time point) by end of study.) | 1428; 8 Hospitals (1428 unique nurses assessed overall (at any time point) by end of study.)
Not Completed | 0; 1 Hospitals | 0; 0 Hospitals
Period: Patient Quality of Care Assessments
Arm/Group | Online ECG Education | Standard Care Then Online ECG Monitoring
Started | 2299; 9 Hospitals (915 unique patients were assessed at 9 hospitals at the initiation of the study.) | 2288; 8 Hospitals (889 unique patients were assessed at 8 hospitals at the initiation of the study.)
Baseline Assessment | 915; 9 Hospitals (915 unique patients, assessed at 9 hospitals.) | 889; 8 Hospitals (889 unique patients, assessed at 8 hospitals.)
15 Months Assessment | 687; 8 Hospitals (687 unique patients, assessed at 8 hospitals.) | 773; 8 Hospitals (773 unique patients, assessed at 8 hospitals.)
30 Months Assessment | 697; 8 Hospitals (697 unique patients, assessed at 8 hospitals.) | 626; 7 Hospitals (626 unique patients, assessed at 7 hospitals.)
Completed | 2299; 8 Hospitals (2299 unique patients assessed overall (at any time point) by end of study.) | 2288; 7 Hospitals (2288 unique patients assessed overall (at any time point) by end of study.)
Not Completed | 0; 1 Hospitals | 0; 1 Hospitals
Period: Patient Outcomes (Hospital Admissions)
Arm/Group | Online ECG Education | Standard Care Then Online ECG Monitoring
Started | 52085; 7 Hospitals (17352 unique patients were assessed at 7 hospitals at the initiation of the study.) | 43799; 6 Hospitals (16459 unique patients were assessed at 6 hospitals at the initiation of the study.)
Baseline Assessment | 17352; 7 Hospitals (17352 unique patients, assessed at 7 hospitals.) | 16549; 6 Hospitals (16549 unique patients, assessed at 6 hospitals.)
15 Months Assessment | 18031; 7 Hospitals (18031 unique patients, assessed at 7 hospitals.) | 14075; 6 Hospitals (14075 unique patients, assessed at 6 hospitals.)
30 Months Assessment | 16702; 7 Hospitals (16702 unique patients, assessed at 7 hospitals.) | 13265; 6 Hospitals (13265 unique patients, assessed at 6 hospitals.)
Completed | 52085; 7 Hospitals (52085 unique patients assessed overall (at any time point) by end of study.) | 43799; 6 Hospitals (43799 unique patients assessed overall (at any time point) by end of study.)
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals

BASELINE CHARACTERISTICS:
Groups:
- Nurses: Nurses on participating units who received education at the time hospital assigned to the standard training or online ECG education training.
- Patients: Patients on participating units on whom quality of care data was obtained.
- Total: Total of all reporting groups
Arm/Group | Nurses | Patients | Total
Number analyzed (Participants) | 3013 | 4587 | 7600
Age, Continuous [Mean (Standard Deviation); unit: years] — Overall age across study groups was not calculated for the different population samples. Population: Age missing for 11 patients.
  years
    number analyzed (Participants) | 3013 | 4576 | 7589
    (all) | 37.53 (11.05) | 65.54 (5.28) | NA (NA) — Overall age across study groups was not calculated for the different population samples.
Sex: Female, Male [Count of Participants; unit: Participants] — Sex missing for 8 patients. Population: Sex missing for 8 patients.
  Participants
    number analyzed (Participants) | 3013 | 4579 | 7592
    Female | 2691 | 1954 | 4645
    Male | 322 | 2625 | 2947
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity missing for 112 patients.
  Participants
    number analyzed (Participants) | 3013 | 4475 | 7488
    Hispanic or Latino | 81 | 226 | 307
    Not Hispanic or Latino | 2932 | 4249 | 7181
    Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants] — Population: Education data not obtained from patients.
  Participants
    number analyzed (Participants) | 3013 | 0 | 3013
    Diploma | 291 |  | 291
    Associate's Degree | 534 |  | 534
    Bachelor's Degree | 1959 |  | 1959
    Master's Degree | 208 |  | 208
    Doctoral Degree | 11 |  | 11
    None of the above | 10 |  | 10
Type of Unit [Count of Participants; unit: Participants] — Population: Unit data not obtained from patients.
  Participants
    number analyzed (Participants) | 3013 | 0 | 3013
    Medicine | 1329 |  | 1329
    Surgery | 830 |  | 830
    Combined | 854 |  | 854

OUTCOME MEASURES:

1. Primary Outcome: Nurses' Knowledge and Skills Related to ECG Monitoring
Description: Participants took a 20-item online test on essentials of ECG monitoring, and arrhythmia, ischemia, and QT interval monitoring. Scores represent the percentage of correct answers. (Test scores range from 0 to 100 with higher scores representing more correct answers)
Time Frame: Baseline, 15 months, 30 months
Population: The overall number of unique nurses assessed at any timepoint. The numbers presented at each time point reflect the number of people assessed at that time point.
Measure: Mean (Standard Deviation); unit: percentage of items correctly answered
Arm/Group | Online ECG Education | Standard Care Then Online ECG Monitoring
Number analyzed (Participants) | 1585 | 1428
percentage of items correctly answered
  Baseline: number analyzed (Participants) | 873 | 866
  Baseline | 49.2 (12.8) | 47.2 (10.8)
  15 Months: number analyzed (Participants) | 1108 | 782
  15 Months | 70.2 (15.5) | 49.4 (11.6)
  30 Months: number analyzed (Participants) | 741 | 926
  30 Months | 59.4 (16.0) | 71.0 (14.3)

2. Secondary Outcome: Quality of Patient Care Related to ECG Monitoring
Description: Percentage of patients with accurate electrode placement, accurate rhythm interpretation, cardiac arrest, cardiac arrest initiated by arrhythmia, appropriate monitoring, telemetry units only, ST-segment monitoring when indicated, and QTc measurement when indicated
Time Frame: Baseline, 15 months, 30 months
Population: The overall number of unique patients assessed at any timepoint. The numbers presented at each time point reflect the number of people assessed at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Online ECG Education | Standard Care Then Online ECG Monitoring
Number analyzed (Participants) | 2299 | 2288
Participants
  Baseline: Right Arm: number analyzed (Participants) | 668 | 691
  Baseline: Right Arm | 579 | 572
  Baseline: Left Arm: number analyzed (Participants) | 668 | 692
  Baseline: Left Arm | 565 | 529
  Baseline: Left Leg: number analyzed (Participants) | 667 | 692
  Baseline: Left Leg | 497 | 494
  Baseline: V Lead: number analyzed (Participants) | 538 | 627
  Baseline: V Lead | 106 | 178
  15 Months: Right Arm: number analyzed (Participants) | 460 | 631
  15 Months: Right Arm | 416 | 520
  15 Months: Left Arm: number analyzed (Participants) | 461 | 630
  15 Months: Left Arm | 411 | 503
  15 Months: Left Leg: number analyzed (Participants) | 457 | 629
  15 Months: Left Leg | 406 | 511
  15 Months: V Lead: number analyzed (Participants) | 386 | 579
  15 Months: V Lead | 229 | 221
  30 Months: Right Arm: number analyzed (Participants) | 475 | 508
  30 Months: Right Arm | 447 | 461
  30 Months: Left Arm: number analyzed (Participants) | 475 | 506
  30 Months: Left Arm | 440 | 457
  30 Months: Left Leg: number analyzed (Participants) | 475 | 505
  30 Months: Left Leg | 435 | 467
  30 Months: V Lead: number analyzed (Participants) | 392 | 449
  30 Months: V Lead | 256 | 280
  Baseline: Accurate Rhythm Interpretation: number analyzed (Participants) | 92 | 75
  Baseline: Accurate Rhythm Interpretation | 75 | 71
  15 Months: Accurate Rhythm Interpretation: number analyzed (Participants) | 74 | 62
  15 Months: Accurate Rhythm Interpretation | 72 | 51
  30 Months: Accurate Rhythm Interpretation: number analyzed (Participants) | 85 | 83
  30 Months: Accurate Rhythm Interpretation | 80 | 81
  Baseline: Cardiac Arrest: number analyzed (Participants) | 915 | 889
  Baseline: Cardiac Arrest | 11 | 5
  15 Months: Cardiac Arrest: number analyzed (Participants) | 685 | 775
  15 Months: Cardiac Arrest | 0 | 10
  30 Months: Cardiac Arrest: number analyzed (Participants) | 697 | 626
  30 Months: Cardiac Arrest | 5 | 2
  Baseline: Cardiac Arrest Initiated by Arrhythmia: number analyzed (Participants) | 915 | 889
  Baseline: Cardiac Arrest Initiated by Arrhythmia | 10 | 4
  15 Months: Cardiac Arrest Initiated by Arrhythmia: number analyzed (Participants) | 685 | 775
  15 Months: Cardiac Arrest Initiated by Arrhythmia | 0 | 9
  30 Months: Cardiac Arrest Initiated by Arrhythmia: number analyzed (Participants) | 695 | 626
  30 Months: Cardiac Arrest Initiated by Arrhythmia | 1 | 1
  Baseline: Appropriate monitoring, telemetry units: number analyzed (Participants) | 685 | 802
  Baseline: Appropriate monitoring, telemetry units | 450 | 543
  15 Months: Appropriate monitoring, telemetry units: number analyzed (Participants) | 549 | 729
  15 Months: Appropriate monitoring, telemetry units | 382 | 433
  30 Months: Appropriate monitoring, telemetry units: number analyzed (Participants) | 665 | 744
  30 Months: Appropriate monitoring, telemetry units | 465 | 536
  Baseline: ST-segment monitoring when indicated: number analyzed (Participants) | 91 | 125
  Baseline: ST-segment monitoring when indicated | 51 | 33
  15 Months: ST-segment monitoring when indicated: number analyzed (Participants) | 89 | 116
  15 Months: ST-segment monitoring when indicated | 60 | 51
  30 Months: ST-segment monitoring when indicated: number analyzed (Participants) | 80 | 85
  30 Months: ST-segment monitoring when indicated | 60 | 38
  Baseline: QTc measurement when indicated: number analyzed (Participants) | 150 | 100
  Baseline: QTc measurement when indicated | 19 | 28
  15 Months: QTc measurement when indicated: number analyzed (Participants) | 162 | 103
  15 Months: QTc measurement when indicated | 83 | 35
  30 Months: QTc measurement when indicated: number analyzed (Participants) | 188 | 147
  30 Months: QTc measurement when indicated | 84 | 51

3. Secondary Outcome: Patient Outcomes
Description: Mortality, in-hospital MI, and not surviving a cardiac arrest were obtained using administrative data and laboratory data (eg, troponin, CK-MB) for all patients. Mortality was defined as death that occurred on one of the participating units. To identify the occurrence of in-hospital MI, laboratory data, timing of procedures, and location of patient at the time of the first blood draw indicating the event were used. Cardiac arrest was defined as an event initiated by an arrhythmia that required immediate intervention and was initiated on a PULSE participating unit. For each qualifying cardiac arrest, it was determined whether the patient survived the event.
Time Frame: Baseline, 15 months, 30 months
Population: The overall number of unique patients reviewed at any timepoint. The numbers presented at each time point reflect the number of people reviewed at that time point for that outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Online ECG Education | Standard Care Then Online ECG Monitoring
Number analyzed (Participants) | 52085 | 43799
Participants
  Baseline: Mortality: number analyzed (Participants) | 12756 | 7802
  Baseline: Mortality | 348 | 218
  Baseline: In-hospital MI: number analyzed (Participants) | 15000 | 13451
  Baseline: In-hospital MI | 355 | 419
  Baseline: Not Survive Cardiac Arrest: number analyzed (Participants) | 38 | 32
  Baseline: Not Survive Cardiac Arrest | 8 | 15
  15 Months: Mortality: number analyzed (Participants) | 14072 | 10180
  15 Months: Mortality | 376 | 194
  15 Months: In-hospital MI: number analyzed (Participants) | 15697 | 14075
  15 Months: In-hospital MI | 303 | 403
  15 Months: Not Survive Cardiac Arrest: number analyzed (Participants) | 44 | 25
  15 Months: Not Survive Cardiac Arrest | 10 | 8
  30 Months: Mortality: number analyzed (Participants) | 13372 | 9234
  30 Months: Mortality | 416 | 223
  30 Months: In-hospital MI: number analyzed (Participants) | 15166 | 13263
  30 Months: In-hospital MI | 225 | 311
  30 Months: Not Survive Cardiac Arrest: number analyzed (Participants) | 48 | 31
  30 Months: Not Survive Cardiac Arrest | 12 | 7

ADVERSE EVENTS:
Description: Only cardiac arrest adverse events were assessed in the Quality of Care patients. Only all-cause mortality (while on a study unit) and Myocardial Infarction adverse events were assessed in the Patient Outcomes patients. These distinctions in data collection methods are why the at risk numbers differ by event and study arm.
Groups:
- Online ECG Education- Patient Outcomes: The intervention consisted of an online ECG monitoring education program (9 mo) and strategies to implement and sustain change in practice (6 mo). Data were collected from both groups at time 2 after group 1 received the intervention. Final data collection occurred at time 3 after group 2 received the intervention. Data collection time points were 15 mo apart. These are Adverse Events reported for the Patient Outcomes groups.
- Standard Care Then Online ECG Monitoring- Patient Outcomes: Hospitals were randomized to administer usual in-service education for nurses for 15 months, then received an online ECG monitoring education program (9 mo) and strategies to implement and sustain change in practice (6 mo). Data were collected from both groups at time 2 after group 1 received the intervention. Final data collection occurred at time 3 after group 2 received the intervention. Data collection time points were 15 mo apart. These are Adverse Events reported for the Patient Outcomes groups.
- Online ECG Education- Quality of Care: The intervention consisted of an online ECG monitoring education program (9 mo) and strategies to implement and sustain change in practice (6 mo). Data were collected from both groups at time 2 after group 1 received the intervention. Final data collection occurred at time 3 after group 2 received the intervention. Data collection time points were 15 mo apart. These are Adverse Events reported for the Patient Quality of Care groups.
- Standard Care Then Online ECG Monitoring- Quality of Care: Hospitals were randomized to administer usual in-service education for nurses for 15 months, then received an online ECG monitoring education program (9 mo) and strategies to implement and sustain change in practice (6 mo). Data were collected from both groups at time 2 after group 1 received the intervention. Final data collection occurred at time 3 after group 2 received the intervention. Data collection time points were 15 mo apart. Patient Quality of Care groups.
Arm/Group | Online ECG Education- Patient Outcomes | Standard Care Then Online ECG Monitoring- Patient Outcomes | Online ECG Education- Quality of Care | Standard Care Then Online ECG Monitoring- Quality of Care
All-Cause Mortality (participants affected / at risk) | 1140/40200 | 635/27216 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 883/52085 | 1045/43799 | 16/2299 | 17/2288
Other Adverse Events (participants affected / at risk) | 0/52085 | 0/43799 | 0/2299 | 0/2288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Online ECG Education- Patient Outcomes (N=52085) | Standard Care Then Online ECG Monitoring- Patient Outcomes (N=43799) | Online ECG Education- Quality of Care (N=2299) | Standard Care Then Online ECG Monitoring- Quality of Care (N=2288)
Myocardial Infarction (MI) (Cardiac disorders) | 883 (883) | 1045 (1045) | 0/0 (0) | 0/0 (0) — Event only assessed in Patient Outcomes groups.
Cardiac Arrest (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 16 (16) | 17 (17) — Event only assessed in Patient Quality of Care groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes